CLINICAL TRIAL: NCT03644706
Title: A Phase 3 Multicenter, Randomized, Double-Blinded, Placebo-Controlled Withdrawal Study Evaluating ADV7103 In Pediatric and Adult Subjects With Distal Renal Tubular Acidosis (dRTA)
Brief Title: Study Evaluating Subjects With Distal Renal Tubular Acidosis
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Research operation issues
Sponsor: Advicenne Pharma (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: B23CS
Record Dates: First submitted 2018-08-22; First posted 2018-08-23 (Actual); Last update posted 2024-03-22 (Actual); Status verified 2024-03

CONDITIONS: Distal Renal Tubular Acidosis
MeSH Terms: conditions — Acidosis, Renal Tubular | interventions — Potassium Citrate; potassium bicarbonate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- ADV7103 (Active Comparator): Patients continue to receive ADV7103 twice a day at their open label dose over 6 days
  Interventions: Drug: ADV7103
- Placebo Comparator (Placebo Comparator): Patients receive matched placebo twice a day until they reach a bicarbonate level of 18mEq/L
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: ADV7103 — Each dose of ADV7103 contains a fixed ratio of 1/3 of ADV7103-CK (potassium citrate) and 2/3 of ADV7103-BK (potassium bicarbonate) based on the mass of active substances. The strength is 6.44 (± 10 %) mEq/g of ADV7103 (alkalinizing power).
  Other Names: Potassium Citrate and Potassium Bicarbonate
  Arms: ADV7103
Drug: Placebo — Placebo is a combination of 2 mm green coated lactose granules and 2 mm white coated lactose granules to be taken by mouth.
  Each dose of placebo contains a fixed ratio of 1/3 of green granules and 2/3 of white granules.
  Arms: Placebo Comparator

SUMMARY:
This is a phase 3, prospective, multicenter, randomized, double-blinded, placebo-controlled withdrawal study comparing the efficacy of ADV7103 versus placebo in preventing the development of metabolic acidosis defined by serum bicarbonate levels in pediatric (6 months to < 18 years of age) and adult (18 to 65 years of age) subjects with primary Distal Renal Tubular Acidosis (dRTA).

DETAILED DESCRIPTION:
The study will target enrolling at least 4 subjects in each of the following age groups: 6 months - 23 months; 2-11 years, and ≥ 12 years. Subjects will be in the study for up to 21 weeks. After screening and enrollment, subjects will participate in an 8-12 week open label period where there dose of ADV7103 will be titrated to effect, then continued for the remainder of the open-label period. Periodic measurements of bicarbonate and potassium levels will be collected during this period. Following the open-label period, subjects will enter a 6-day randomized withdrawal period. A follow-up period up to four weeks on re-established therapy completes the trial. Subjects can elect to return to their previous standard of care regimen after completing the withdrawal period or will have the opportunity to subsequently enter an open-label extension study.

ELIGIBILITY:
Inclusion Criteria:

1. Female or male subjects ≥ 6 months of age and ≤ 65 years of age at time of consent;
2. Subject presents with a previous diagnosis of primary dRTA of at least 4 months duration for subjects < 12 years of age, and at least one year for those ≥ 12 years of age, based on documented history of non-anion gap, hyperchloremic, hypokalemic metabolic acidosis;
3. Subject requires ≥ 0.9 mEq/kg/day of alkali therapy to maintain serum bicarbonate levels above the LLN for the laboratory providing results;
4. Subject or parent/guardian is willing and able to understand and sign informed consent and willing to comply with protocol instructions; child assent when appropriate; and
5. Heterosexually active female subjects of childbearing potential and non-sterilized males must use at least one of the following acceptable birth control methods from informed consent through 7 days after the last dose of study product:

   1. Double-barrier methods of contraception: condom or occlusive cap (diaphragm or cervical/vault caps) with spermicidal foam/gel/film/cream/suppository)
   2. Established use of oral, injectable, or implanted hormonal methods of contraception
   3. Placement of an intrauterine device or intrauterine system
   4. Abstinence Females of childbearing potential are those who have reached the onset of menarche (or 8 years of age, whichever comes first) and are not postmenopausal (≥ 1 year without menses prior to Visit 1), surgically sterile, or status post hysterectomy (≥ 1 month prior to Visit 1). From informed consent through 7 days after the last dose of study product, female subjects must agree to refrain from egg donation and male subjects must agree to refrain from sperm donation.

Exclusion Criteria:

1. Female subject who is pregnant or lactating or has plans for pregnancy during the study;
2. Subject has evidence of proximal tubule dysfunction (eg, hypophosphatemia, low serum uric acid, glycosuria, or amino aciduria);
3. Subject presents with another diagnosed condition as a potential etiology for her/his dRTA (eg, systemic lupus erythematosus, Sjogren's syndrome), in the opinion of the Investigator;
4. Subject requires therapy with potassium sparing diuretics, angiotensin converting enzyme inhibitors, angiotensin II receptor blockers, trimethoprim, drospirenone and other progestins, nephrotoxic antibiotics, penicillins, tacrolimus, or medications known to delay gastric emptying or otherwise interfere with absorption of study product;
5. Subject has evidence of obstructive uropathy or other findings on renal ultrasound associated with Visit 1 expected to require intervention during the course of the study, in the opinion of the Investigator;
6. Subject has any of the following laboratory abnormalities associated with Visit 1:

   1. AST and/or ALT > 1.5x upper limit of normal (ULN)
   2. Serum potassium > 5.0 mEq/L or <3.0 mEq/L or hypokalemia accompanied by clinical symptoms (eg, muscle cramps) or significant ECG changes (eg T wave depression, U wave elevation)
   3. Estimated glomerular filtration rate (eGFR) < 60 mL/min/1.73 m2 (according to the Modified Schwartz formula for children [<12years of age] and Chronic Kidney Disease - Epidemiology Collaboration [CKD-EPI] equation for adolescents and adults [≥12 years of age])
   4. Total bilirubin > ULN, except with known Gilbert's disease or in patients with dRTA and known hemolytic anemia due to a defect in SLC4A1.
7. Subject has been hospitalized or had outpatient surgery (other than minor skin and dRTA disease-related procedures or ear tube placement) in the past 6 months or is planning surgery in the next 6 months;
8. In the opinion of the Investigator, the subject has a major medical or psychiatric condition (eg, significant cardiac disease, schizophrenia) or an unstable condition (eg, uncontrolled hypertension, asthma, diabetes, hypercholesterolemia, or cardiac disease) that would potentially interfere with the subject safely completing the study;
9. In the opinion of the Investigator, the subject has a history of difficulty taking oral medication and/or conditions that may hinder absorption of the study drug (eg, any difficulty of swallowing, malabsorption, delayed gastric emptying, esophageal compression, intestinal obstruction, or other chronic gastrointestinal disease);
10. Self-reported or parent/guardian reported alcohol abuse or drug abuse within the past 12 months;
11. Subject is a solid organ or bone marrow transplant recipient;
12. Subject has a history of malignancy within 5 years prior to Visit 1, except for localized skin or cervical carcinoma; or
13. Subject is known to have allergy or intolerance to any ADV7103 or placebo constituents.

Ages: 6 Months to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2021-09-20 (Actual); Primary Completion 2023-12-20 (Actual); Study Completion 2023-12-20 (Actual)

PRIMARY OUTCOMES:
Mean change in blood bicarbonate levels | 6 days
  Compare the efficacy of ADV7103 versus placebo in preventing metabolic acidosis, defined as 2 consecutive serum bicarbonate levels < 18 mEq/L for subjects ≥ 4 years old and < 17 mEq/L for subjects < 4 years old, during the Withdrawal Period

CONTACTS AND LOCATIONS:
Overall Officials: Laurence Greenbaum, MD, Ph.D., Principal Investigator — Emory University
Locations (8):
- United States (6):
  - Children's Hospital Colorado, Aurora, Colorado
  - University of South Florida Pediatric Infectious Disease, Tampa, Florida
  - Emory Children's Center, Atlanta, Georgia
  - J.W. Riley Hospital for Children/Indiana University, Indianapolis, Indiana
  - Montefiore Medical Center, The Bronx, New York
  - The Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
- Canada (2):
  - University of Alberta, Edmonton, Alberta
  - The Hospital for Sick Children, Toronto, Ontario

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Patient education — https://www.kidney.org/atoz/content/dRTA
- See also: Company website — http://advicenne.com/